CLINICAL TRIAL: NCT02951182
Title: A Phase 2, Randomized, Double-blind, Controlled Study to Evaluate the Safety and Efficacy of VX-440 Combination Therapy in Subjects Aged 12 Years and Older With Cystic Fibrosis
Brief Title: A Study Evaluating the Safety and Efficacy of VX-440 Combination Therapy in Subjects With Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX15-440-101; 2016-000454-36 (EudraCT Number)
Record Dates: First submitted 2016-10-26; First posted 2016-11-01 (Estimated); Results first posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — tezacaftor; ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Part 1: Placebo - Cohort 1A and 1B Combined (Placebo Comparator): Participants received placebo matched to VX-440/TEZ/IVA as triple combination for 4 weeks.
  Interventions: Drug: Matched Placebo
- Part 1 Cohort 1A: Triple Combination (TC) (Experimental): Participants received VX-440 200 milligram (mg) every 12 hours (q12h)/TEZ 100 mg once daily (qd)/IVA 150 mg q12h as triple combination for 4 weeks.
  Interventions: Drug: TEZ; Drug: IVA; Drug: VX-440
- Part 1 Cohort 1B: TC Low Dose (Experimental): Participants received VX-440 200 mg q12h/TEZ 50 mg q12h/IVA 150 mg q12h as triple combination for 4 weeks.
  Interventions: Drug: TEZ; Drug: IVA; Drug: VX-440
- Part 1 Cohort 1B: TC High Dose (Experimental): Participants received VX-440 600 mg q12h/TEZ 50 mg q12h/IVA 300 mg q12h as triple combination for 4 weeks.
  Interventions: Drug: TEZ; Drug: IVA; Drug: VX-440
- Part 2: TEZ/IVA (Active Comparator): Following a 4-week run-in period on TEZ 100 mg qd/IVA150 mg q12h, participants received placebo matched to VX-440 and TEZ 50 mg q12h/IVA 300 mg q12h for 4 weeks in treatment period and TEZ 100 mg qd/IVA150 mg q12h for 4 weeks in washout period.
  Interventions: Drug: TEZ; Drug: IVA; Drug: Matched Placebo
- Part 2: TC-2 (Experimental): Following a 4-week run-in period on TEZ 100 mg qd/IVA150 mg q12h, participants received VX-440 600 mg q12h/ TEZ 50 mg q12h/IVA 300 mg q12h for 4 weeks for 4 weeks in treatment period and TEZ 100 mg qd/IVA150 mg q12h for 4 weeks in washout period.
  Interventions: Drug: TEZ; Drug: IVA; Drug: VX-440

INTERVENTIONS:
Drug: TEZ
  Other Names: tezacaftor; VX-661
  Arms: Part 1 Cohort 1A: Triple Combination (TC); Part 1 Cohort 1B: TC High Dose; Part 1 Cohort 1B: TC Low Dose; Part 2: TC-2; Part 2: TEZ/IVA
Drug: IVA
  Other Names: ivacaftor; VX-770
  Arms: Part 1 Cohort 1A: Triple Combination (TC); Part 1 Cohort 1B: TC High Dose; Part 1 Cohort 1B: TC Low Dose; Part 2: TC-2; Part 2: TEZ/IVA
Drug: VX-440
  Arms: Part 1 Cohort 1A: Triple Combination (TC); Part 1 Cohort 1B: TC High Dose; Part 1 Cohort 1B: TC Low Dose; Part 2: TC-2
Drug: Matched Placebo
  Arms: Part 1: Placebo - Cohort 1A and 1B Combined; Part 2: TEZ/IVA

SUMMARY:
This is a Phase 2, randomized, double-blind, placebo- and active-controlled, parallel group, multicenter study to evaluate the safety, tolerability, and efficacy of VX-440 in dual and triple combination with tezacaftor (TEZ; VX-661) and ivacaftor (IVA; VX-770) in subjects with cystic fibrosis (CF) who are homozygous for the F508del mutation of the CF transmembrane conductance regulator (CFTR) gene (F508del/F508del), or who are heterozygous for the F508del mutation and a minimal function (MF) CFTR mutation not likely to respond to TEZ and/or IVA therapy (F508del/MF).

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to comply with scheduled visits, treatment plan, study restrictions, laboratory tests, contraceptive guidelines, and other study procedures.
* To prevent pregnancy, female participants of childbearing potential and their male partners will be required to use pre-specified, highly effective methods of non-hormonal contraception. Male participants with female partners of childbearing potential will be required to use a condom.
* Body weight ≥35 kg.
* Sweat chloride value ≥60 mmol/L from test results obtained during screening.
* Subjects must have an eligible CFTR genotype:

  * Heterozygous for F508del and a minimal function (MF) mutation known or predicted not to be responsive to TEZ and/or IVA.
  * Homozygous for F508del
* Subjects must have an FEV1 ≥40% and ≤90% of predicted normal for age, sex, and height at the Screening Visit
* Stable CF disease as judged by the investigator.
* Willing to remain on a stable CF medication regimen through the planned end of treatment or, if applicable, the Safety Follow up Visit.

Exclusion Criteria:

* History of any comorbidity that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject.
* History of cirrhosis with portal hypertension.
* Risk factors for Torsade de Pointes
* History of hemolysis.
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency assessed at Screening.
* Clinically significant abnormal laboratory values at screening
* An acute upper or lower respiratory infection, pulmonary exacerbation, or changes in therapy for pulmonary disease within 28 days before the first dose of study drug.
* Lung infection with organisms associated with a more rapid decline in pulmonary status
* An acute illness not related to CF within 14 days before the first dose of study drug
* A standard digital ECG demonstrating QTc >450 msec at screening.
* History of solid organ or hematological transplantation.
* History or evidence of cataract or lens opacity determined to be clinically significant by the ophthalmologist or optometrist based on the ophthalmologic examination during the Screening Period.
* History of alcohol or drug abuse in the past year, including but not limited to, cannabis, cocaine, and opiates, as deemed by the investigator.
* Ongoing or prior participation in an investigational drug study, with certain exceptions. (e.g., ongoing participation in NCT02565914)
* Use of commercially available CFTR modulator (e.g., Kalydeco, Orkambi) within 14 days before screening (applies only to the Heterozygous F508del/MF cohorts; does not apply to the Homozygous F508del/F508del Cohort).
* Pregnant or nursing females: Females of childbearing potential must have a negative pregnancy test at screening and Day 1.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (40):
- United States (22):
  - The Arizona Board of Regents on behalf of the University of Arizona, Tucson, Arizona
  - Stanford University, Palo Alto, California
  - University of California, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - Joe Di Maggio Cystic Fibrosis & Pulmonary Center, Hollywood, Florida
  - Central Florida Pulmonary Group, Orlando, Florida
  - St. Luke's CF Center of Idaho, Boise, Idaho
  - Cystic Fibrosis Center of Chicago, Glenview, Illinois
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital Cystic Fibrosis Center, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - New York Medical College, Hawthorne, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Columbia University Medical Center, New York, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - Respiratory Diseases of Children and Adolescents, Oklahoma City, Oklahoma
  - UPMC OSPARS Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Sanford Children's Specialty Clinic Sanford Research USD, Sioux Falls, South Dakota
  - The University of Texas Southwestern Center, Dallas, Texas
  - Children's Hospital of the Kings Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
- Australia (3):
  - Royal Adelaide Hospital, Adelaide
  - Prince Charles Hospital, Chermside
  - John Hunter Hospital & Hunter Medical Research Institute, New Lambton Heights
- Medizinische Universitat Innsbruck, Innsbruck, Austria
- Belgium (2):
  - Universitair Ziekenhuis Brussel, Brussels
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
- Canada (2):
  - St. Paul's Hopsital, Vancouver, British Columbia
  - St. Michael's Hospital, Toronto, Ontario
- Juliane Marie Center, Righospitalet, Copenhagen, Denmark
- Germany (3):
  - University Hospital Cologne, Cologne
  - Mukeviszidose-Zentrum am Universtitatsklinikum Jena, Jena
  - Pneumologische Praxis Pasing, München
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy
- Spain (2):
  - Hospital Universitari Vall d´Hebron Servicio de Broncoscopia, Barcelona
  - Hospital Universitario Virgen del Rocio, Seville
- United Kingdom (3):
  - Heart of England NHS Foundation Trust, Birmingham
  - Royal Brompton & Harefield NHS Foundation Trust, Royal Brompton Hospital, London
  - Southampton University Hospitals NHS Foundation Trust, Southampton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 74 participants enrolled (47 participants in Part 1 and 27 participants in Part 2), 1 participant in Part 2 discontinued in the Run-in Period because continuation criteria were not met and was not randomized in the Treatment Period. Therefore, only 73 participants are included in the results below.
Pre-assignment Details: Four parts were originally planned for the study; only Parts 1 and 2 were conducted. Part 3 was removed in protocol Version 2.0. Part 4 was not conducted at the Sponsor's discretion.
Groups:
- Part 1: Placebo - Cohort 1A and 1B Combined: Participants received placebo matched to VX-440/tezacaftor (TEZ; VX-661)/ivacaftor (IVA, VX-770) as triple combination for 4 weeks.
Period: Overall Study
Arm/Group | Part 1: Placebo - Cohort 1A and 1B Combined | Part 1 Cohort 1A: Triple Combination (TC) | Part 1 Cohort 1B: TC Low Dose | Part 1 Cohort 1B: TC High Dose | Part 2: TEZ/IVA | Part 2: TC-2
Started | 11 | 9 | 9 | 18 | 6 | 20
Completed | 11 | 9 | 9 | 18 | 6 | 20
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1 Cohort 1A: Triple Combination (TC): Participants received VX-440 200 mg q12h/TEZ 100 mg qd/IVA 150 mg q12h as triple combination for 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Part 1: Placebo - Cohort 1A and 1B Combined | Part 1 Cohort 1A: Triple Combination (TC) | Part 1 Cohort 1B: TC Low Dose | Part 1 Cohort 1B: TC High Dose | Part 2: TEZ/IVA | Part 2: TC-2 | Total
Number analyzed (Participants) | 11 | 9 | 9 | 18 | 6 | 20 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 9 | 18 | 6 | 20 | 73
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3 | 1 | 0 | 4 | 11
  Male | 9 | 8 | 6 | 17 | 6 | 16 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 0 | 1 | 3
  Not Hispanic or Latino | 10 | 9 | 8 | 17 | 6 | 18 | 68
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 10 | 9 | 9 | 18 | 6 | 20 | 72
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability as Assessed by Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: From first dose of Study Drug in the Treatment Period through Safety Follow-up Visit (Up to Day 57 for Part 1 and Day 85 for Part 2)
Population: Safety Set included all participants who received at least 1 dose of study drug in the Treatment Period.
Measure: Number; unit: participants
Arm/Group | Part 1: Placebo - Cohort 1A and 1B Combined | Part 1 Cohort 1A: Triple Combination (TC) | Part 1 Cohort 1B: TC Low Dose | Part 1 Cohort 1B: TC High Dose | Part 2: TEZ/IVA | Part 2: TC-2
Number analyzed (Participants) | 11 | 9 | 9 | 18 | 6 | 20
participants
  Participants with AEs | 9 | 9 | 9 | 15 | 6 | 15
  Participants with SAEs | 0 | 0 | 0 | 2 | 2 | 1

2. Primary Outcome: Absolute Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline through Day 29
Population: Full Analysis Set (FAS) included all randomized participants who have received at least 1 dose of study drug in the Treatment Period. As per pre-specified planned analysis, reporting group "Part 1 Cohort 1A: TC" and "Part 1 Cohort 1B: TC Low Dose" were pooled for the purpose of efficacy analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage points
Groups:
- Part 1: TC-1A/ TC-1B-low Pooled: All participants pooled together for Part 1: TC-1A arm and Part 1: TC-1B low dose arm.
Arm/Group | Part 1: Placebo - Cohort 1A and 1B Combined | Part 1: TC-1A/ TC-1B-low Pooled | Part 1 Cohort 1B: TC High Dose | Part 2: TEZ/IVA | Part 2: TC-2
Number analyzed (Participants) | 11 | 18 | 18 | 6 | 20
percentage points | 1.4 [-2.7 to 5.5] | 10.0 [6.9 to 13.2] | 12.0 [8.8 to 15.2] | -2.5 [-7.2 to 2.2] | 9.5 [6.9 to 12.2]
Statistical Analysis 1: Comparison: Part 1: Placebo - Cohort 1A and 1B Combined vs Part 1: TC-1A/ TC-1B-low Pooled; Test type: Superiority; p = 0.0016, Mixed-effects Model for Repeated Measure; Least Squares (LS) Mean Difference = 8.6, 95% CI 2-sided [3.5 to 13.8]
Statistical Analysis 2: Comparison: Part 1: Placebo - Cohort 1A and 1B Combined vs Part 1 Cohort 1B: TC High Dose; Test type: Superiority; p = 0.0001, Mixed-effects Model for Repeated Measure; Least Squares (LS) Mean Difference = 10.6, 95% CI 2-sided [5.5 to 15.8]
Statistical Analysis 3: Comparison: Part 2: TEZ/IVA vs Part 2: TC-2; Test type: Superiority; p = 0.0001, Mixed-effects Model for Repeated Measure; Least Squares (LS) Mean Difference = 12.0, 95% CI 2-sided [6.7 to 17.4]

3. Secondary Outcome: Absolute Change in Sweat Chloride Concentrations
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline through Day 29
Population: FAS. As per pre-specified planned analysis, reporting group "Part 1 Cohort 1A: TC" and "Part 1 Cohort 1B: TC Low Dose" were pooled for the purpose of efficacy analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimole per liter (mmol/L)
Arm/Group | Part 1: Placebo - Cohort 1A and 1B Combined | Part 1: TC-1A/ TC-1B-low Pooled | Part 1 Cohort 1B: TC High Dose | Part 2: TEZ/IVA | Part 2: TC-2
Number analyzed (Participants) | 11 | 18 | 18 | 6 | 20
millimole per liter (mmol/L) | 1.6 [-6.2 to 9.4] | -20.7 [-26.6 to -14.7] | -33.1 [-39.1 to -27.1] | 2.1 [-10.9 to 15.1] | -31.3 [-38.6 to -24.1]
Statistical Analysis 1: Comparison: Part 1: Placebo - Cohort 1A and 1B Combined vs Part 1: TC-1A/ TC-1B-low Pooled; Test type: Superiority; Least Squares (LS) Mean Difference = -22.3, 95% CI 2-sided [-32.1 to -12.4]
Statistical Analysis 2: Comparison: Part 1: Placebo - Cohort 1A and 1B Combined vs Part 1 Cohort 1B: TC High Dose; Test type: Superiority; Least Squares (LS) Mean Difference = -34.7, 95% CI 2-sided [-44.7 to -24.8]
Statistical Analysis 3: Comparison: Part 2: TEZ/IVA vs Part 2: TC-2; Test type: Superiority; Least Squares (LS) Mean Difference = -33.4, 95% CI 2-sided [-48.5 to -18.3]

4. Secondary Outcome: Relative Change in ppFEV1
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline through Day 29
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Part 1: Placebo - Cohort 1A and 1B Combined | Part 1: TC-1A/ TC-1B-low Pooled | Part 1 Cohort 1B: TC High Dose | Part 2: TEZ/IVA | Part 2: TC-2
Number analyzed (Participants) | 11 | 18 | 18 | 6 | 20
percent change | 2.6 [-4.9 to 10.0] | 17.3 [11.5 to 23.2] | 21.7 [15.9 to 27.5] | -3.4 [-11.4 to 4.6] | 16.6 [12.1 to 21.1]
Statistical Analysis 1: Comparison: Part 1: Placebo - Cohort 1A and 1B Combined vs Part 1: TC-1A/ TC-1B-low Pooled; Test type: Superiority; Least Squares (LS) Mean Difference = 14.8, 95% CI 2-sided [5.3 to 24.2]
Statistical Analysis 2: Comparison: Part 1: Placebo - Cohort 1A and 1B Combined vs Part 1 Cohort 1B: TC High Dose; Test type: Superiority; Least Squares (LS) Mean Difference = 19.1, 95% CI 2-sided [9.7 to 28.6]
Statistical Analysis 3: Comparison: Part 2: TEZ/IVA vs Part 2: TC-2; Test type: Superiority; Least Squares (LS) Mean Difference = 20.0, 95% CI 2-sided [10.8 to 29.1]

5. Secondary Outcome: Absolute Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms, score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life.
Time Frame: From Baseline at Day 29
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Part 1: Placebo - Cohort 1A and 1B Combined | Part 1: TC-1A/ TC-1B-low Pooled | Part 1 Cohort 1B: TC High Dose | Part 2: TEZ/IVA | Part 2: TC-2
Number analyzed (Participants) | 11 | 18 | 18 | 6 | 20
units on a scale | 2.2 [-6.2 to 10.6] | 18.3 [11.7 to 24.9] | 20.7 [14.2 to 27.1] | -7.8 [-14.8 to -0.8] | 12.3 [8.7 to 16.0]
Statistical Analysis 1: Comparison: Part 1: Placebo - Cohort 1A and 1B Combined vs Part 1: TC-1A/ TC-1B-low Pooled; Test type: Superiority; Least Squares (LS) Mean Difference = 16.1, 95% CI 2-sided [5.4 to 26.8]
Statistical Analysis 2: Comparison: Part 1: Placebo - Cohort 1A and 1B Combined vs Part 1 Cohort 1B: TC High Dose; Test type: Superiority; Least Squares (LS) Mean Difference = 18.5, 95% CI 2-sided [7.9 to 29.1]
Statistical Analysis 3: Comparison: Part 2: TEZ/IVA vs Part 2: TC-2; Test type: Superiority; Least Squares (LS) Mean Difference = 20.2, 95% CI 2-sided [11.9 to 28.4]

6. Secondary Outcome: Pre-dose Plasma Concentration (Ctrough) of VX-440, TEZ, M1-TEZ, IVA and M1-IVA
Time Frame: Predose at Day 8, Day 15 and Day 29
Population: Pharmacokinetic Set (PK) included all participants who have received at least 1 dose of study drug in Treatment Period. Here "Number Analyzed" signifies those participants who were evaluable at specified time points. Day 8 assessment was planned for only TC-1A arm and VX-440 Ctrough category was not applicable for TEZ/IVA arm.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part 1 Cohort 1A: Triple Combination (TC) | Part 1 Cohort 1B: TC Low Dose | Part 1 Cohort 1B: TC High Dose | Part 2: TEZ/IVA | Part 2: TC-2
Number analyzed (Participants) | 9 | 9 | 18 | 6 | 19
nanogram per milliliter (ng/mL)
  VX-440: Day 8: number analyzed (Participants) | 9 | 0 | 0 | 0 | 0
  VX-440: Day 8 | 1670 (1910) |  |  |  |
  VX-440: Day 15: number analyzed (Participants) | 9 | 8 | 16 | 0 | 18
  VX-440: Day 15 | 1840 (1460) | 1120 (707) | 8540 (6850) |  | 12900 (9940)
  VX-440: Day 29: number analyzed (Participants) | 9 | 9 | 17 | 0 | 17
  VX-440: Day 29 | 1090 (1010) | 1440 (1870) | 6650 (3500) |  | 10300 (7340)
  TEZ: Day 8: number analyzed (Participants) | 8 | 0 | 0 | 0 | 0
  TEZ: Day 8 | 810 (323) |  |  |  |
  TEZ: Day 15: number analyzed (Participants) | 9 | 8 | 16 | 6 | 18
  TEZ: Day 15 | 749 (271) | 1070 (422) | 928 (558) | 2240 (1010) | 1250 (837)
  TEZ: Day 29: number analyzed (Participants) | 9 | 9 | 17 | 6 | 17
  TEZ: Day 29 | 761 (320) | 1040 (659) | 846 (514) | 1420 (565) | 893 (579)
  M1-TEZ: Day 8: number analyzed (Participants) | 8 | 0 | 0 | 0 | 0
  M1-TEZ: Day 8 | 3160 (645) |  |  |  |
  M1-TEZ: Day 15: number analyzed (Participants) | 9 | 8 | 16 | 6 | 18
  M1-TEZ: Day 15 | 3490 (486) | 4610 (1170) | 3400 (1270) | 4640 (1730) | 3940 (1200)
  M1-TEZ: Day 29: number analyzed (Participants) | 9 | 9 | 17 | 6 | 17
  M1-TEZ: Day 29 | 3560 (378) | 4180 (1950) | 3050 (1260) | 4060 (1560) | 3280 (1230)
  IVA: Day 8: number analyzed (Participants) | 8 | 0 | 0 | 0 | 0
  IVA: Day 8 | 281 (167) |  |  |  |
  IVA: Day 15: number analyzed (Participants) | 9 | 8 | 16 | 6 | 18
  IVA: Day 15 | 245 (92.7) | 192 (97.0) | 233 (149) | 1040 (352) | 380 (312)
  IVA: Day 29: number analyzed (Participants) | 9 | 9 | 17 | 6 | 17
  IVA: Day 29 | 209 (112) | 164 (108) | 219 (139) | 902 (344) | 290 (263)
  M1-IVA: Day 8: number analyzed (Participants) | 8 | 0 | 0 | 0 | 0
  M1-IVA: Day 8 | 795 (327) |  |  |  |
  M1-IVA: Day 15: number analyzed (Participants) | 9 | 8 | 16 | 6 | 18
  M1-IVA: Day 15 | 854 (427) | 566 (245) | 850 (546) | 1640 (218) | 1220 (796)
  M1-IVA: Day 29: number analyzed (Participants) | 9 | 9 | 17 | 6 | 17
  M1-IVA: Day 29 | 702 (372) | 520 (338) | 792 (466) | 1580 (764) | 1080 (732)

ADVERSE EVENTS:
Time Frame: From first dose of Study Drug in the Treatment Period through Safety Follow-up Visit (Up to Day 57 for Part 1 and Day 85 for Part 2)
Groups:
- Part 1 Cohort 1A: Triple Combination (TC): Participants received VX-440 200 mg q12/TEZ 100 mg qd/IVA 150 mg q12h as triple combination for 4 weeks.
Arm/Group | Part 1: Placebo - Cohort 1A and 1B Combined | Part 1 Cohort 1A: Triple Combination (TC) | Part 1 Cohort 1B: TC Low Dose | Part 1 Cohort 1B: TC High Dose | Part 2: TEZ/IVA | Part 2: TC-2
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/9 | 0/9 | 0/18 | 0/6 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9 | 0/9 | 2/18 | 2/6 | 1/20
Other Adverse Events (participants affected / at risk) | 9/11 | 9/9 | 9/9 | 15/18 | 5/6 | 15/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo - Cohort 1A and 1B Combined (N=11) | Part 1 Cohort 1A: Triple Combination (TC) (N=9) | Part 1 Cohort 1B: TC Low Dose (N=9) | Part 1 Cohort 1B: TC High Dose (N=18) | Part 2: TEZ/IVA (N=6) | Part 2: TC-2 (N=20)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1
Adjustment disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo - Cohort 1A and 1B Combined (N=11) | Part 1 Cohort 1A: Triple Combination (TC) (N=9) | Part 1 Cohort 1B: TC Low Dose (N=9) | Part 1 Cohort 1B: TC High Dose (N=18) | Part 2: TEZ/IVA (N=6) | Part 2: TC-2 (N=20)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 1 | 1 | 0 | 5
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 1 | 1 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 2 | 6 | 0 | 2 | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 2 | 2 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 2 | 0 | 2
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 2 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 2 | 0 | 1
Blood urine present (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood bicarbonate decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood bilirubin unconjugated increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood chloride increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Crystal urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Lipase decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Monocyte count increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary function test decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 2 | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Abnormal faeces (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Faeces pale (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Tendon discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anaesthetic complication neurological (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 2 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mood swings (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Testicular cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-06-12): https://cdn.clinicaltrials.gov/large-docs/82/NCT02951182/SAP_000.pdf
  • Study Protocol (2016-09-16): https://cdn.clinicaltrials.gov/large-docs/82/NCT02951182/Prot_001.pdf